CLINICAL TRIAL: NCT01199601
Title: Pilot Educational Intervention to Determine Effect of Intrapartum Testing and Concentrated Postpartum Counseling on Birth Spacing, Breastfeeding, and Infant Vaccination Completion in a Kabul Urban Population.
Brief Title: Blood-borne Infection Screening in an Afghan Antenatal Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAD1784; 7K01TW007408-04 (NIH)
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Viral Hepatitis B; Contraception; Breast Feeding, Exclusive; Effects of; Lack of Care of Infants
MeSH Terms: conditions — Hepatitis B; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concentrated postpartum counseling (Experimental): Women randomized to receiving concentrated postpartum counseling from the retrained provider.
  Interventions: Behavioral: Concentrated postpartum counseling
- Routine postpartum counseling (No Intervention): Women receiving intra-partum testing and post-partum counseling from existing cadres of hospital providers at standard of care.

INTERVENTIONS:
Behavioral: Concentrated postpartum counseling — Intrapartum testing and concentrated postpartum counseling for the female patient from a retrained provider focusing on correct breastfeeding practices, postpartum contraception, and infant vaccination.
  Arms: Concentrated postpartum counseling

SUMMARY:
Baseline information indicates there are measurable levels of hepatitis B SAg and low utilization of postpartum contraception, correct breastfeeding practices, or adherence to infant vaccination schedules in Kabul, Afghanistan. This intervention will randomize hospitals to assess the following aims:

Aim 1: To determine whether the re-training and assignment of health care providers dedicated to intrapartum rapid testing and post-partum counseling will positively impact maternal and neonatal health indicators as compared to utilization of existing health providers for these services among women delivering in publish health maternity hospitals in Kabul, Afghanistan.

Aim 2: To assess whether patients randomized to the intervention and their spouses perceive value in concentrated post-partum counseling.

Aim 3: To investigate whether an intervention providing immediate post-partum provision of a long-acting family planning method would be feasible and acceptable to both men and women in Kabul, Afghanistan.

DETAILED DESCRIPTION:
Outcomes are assessed through questionnaire responses and inspection of vaccination cards at six month intervals by trained study staff through one year total study time. Differences between groups will be assessed with generalized linear mixed modeling. Information obtained to address Aim 3 will be gathered at the 12 month follow-up and analyzed with simple proportions and Chi-square test to assess differences between sexes and other socioeconomic indicators.

ELIGIBILITY:
Inclusion Criteria:

* admitted for obstetric care
* Dari or Pashto speaking
* not previously participated in the study
* in medically stable condition
* accompanied by and have approval of a spouse
* able to provide informed consent

Male participants must be the confirmed spouses of the female participants, have a working telephone, and able to provide informed consent.

Exclusion Criteria:

* medically unstable or imminently delivering (complete cervical dilation)
* husband unavailable or does not approve participation
* unable to provide consent

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1291 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Todd, MD, Principal Investigator — Columbia University
Locations (1):
- Maternity Hospitals, Kabul, Afghanistan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women in active labor able to provide consent recruited by random number designation at four Kabul public maternity hospitals following admission. Recruitment occurred from June 2008 through January 2009.
Groups:
- Counseling Existing Providers: Women receiving intra-partum testing and the usual post-partum counseling from existing hospital providers of same professional cadre as intervention group.
  Intrapartum, postpartum counseling : Intrapartum testing and routine counseling package provided by study.
- Counseling, Retrained Provider: Women randomized to receiving intra-partum testing and concentrated counseling from the retrained provider (intervention)
  Intrapartum, postpartum counseling : Intrapartum testing and concentrated counseling from a retrained provider
Period: Overall Study
Arm/Group | Counseling Existing Providers | Counseling, Retrained Provider
Started | 422 (Control Group) | 422 (Intervention Group)
Completed | 353 | 344
Not Completed | 69 | 78
Not completed — Lost to Follow-up | 47 | 66
Not completed — Withdrawal by Subject | 15 | 3
Not completed — Insecurity prevented staff interviewing. | 7 | 9

BASELINE CHARACTERISTICS:
Population: The 1291 reflects the husbands interviewed at 12 months (n=447). The husbands were not analyzed as part of the RCT.
Groups:
- Counseling Existing Providers: Women receiving intra-partum testing and the usual post-partum counseling from existing hospital providers (control group) .
  Intrapartum, postpartum counseling : Intrapartum testing and routine counseling.
- Counseling, Retrained Provider: Women randomized to receiving intra-partum testing and concentrated counseling from the retrained provider (intervention group).
  Intrapartum, postpartum counseling : Intrapartum testing and concentrated counseling from a retrained provider
- Total: Total of all reporting groups
Arm/Group | Counseling Existing Providers | Counseling, Retrained Provider | Total
Number analyzed (Participants) | 422 | 422 | 844
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 31 | 65
  Between 18 and 65 years | 388 | 391 | 779
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (5.6) | 24.8 (5.5) | 24.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 422 | 422 | 844
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Afghanistan | 422 | 422 | 844

OUTCOME MEASURES:

1. Primary Outcome: Utilization of Postpartum Contraception
Description: Determine whether the re-training and assignment of healthcare providers dedicated to intrapartum rapid testing and intensive post-partum counseling will positively impact postpartum contraceptive use as compared to any counseling provided by existing health providers for these services among women delivering in public health maternity hospitals in Kabul, Afghanistan.
Time Frame: 12 months
Population: Participants included in analysis were those completing the 6 and 12 month follow-up visits.
Measure: Number; unit: participants
Groups:
- Counseling Existing Providers: Women receiving intra-partum testing and the usual post-partum counseling from re-trained hospital providers of same professional cadre as control group.
  Intrapartum, postpartum counseling : Intrapartum testing and concentrated counseling package provided by study.
- Counseling, Retrained Provider: Women randomized to receiving intra-partum testing and concentrated counseling from the retrained provider
  Intrapartum, postpartum counseling : Intrapartum testing and concentrated counseling from a retrained provider
Arm/Group | Counseling Existing Providers | Counseling, Retrained Provider
Number analyzed (Participants) | 353 | 344
participants | 199 | 213
Statistical Analysis 1: Comparison: Counseling Existing Providers vs Counseling, Retrained Provider; Outcomes were assessed by crude and adjusted risk ratios with log-binomial generalized linear models; Test type: Superiority or Other; p < 0.05, Regression, Linear; Information provided for crude analysis results; adjustment for significant baseline differences between groups did not change results substantially; Incidence Rate Ratio = 1.12, 95% CI 2-sided [1.02 to 1.23], Standard Deviation .05

2. Secondary Outcome: Correct Breastfeeding Practices to 1 Year
Description: Assess whether patients randomized to the intervention exhibit correct breastfeeding practices (a composite variable in which exclusive breastfeeding occurs to 6 months and continued complementary breastfeeding continues to 12 months) after receiving concentrated postpartum counseling compared to women receiving standard of care.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Counseling Existing Providers | Counseling, Retrained Provider
Number analyzed (Participants) | 353 | 344
participants | 198 | 240
Statistical Analysis 1: Comparison: Counseling Existing Providers vs Counseling, Retrained Provider; Test type: Superiority or Other; p < 0.05, Regression, Linear; Outcomes were assessed by crude and adjusted risk ratios with log-binomial generalized linear models; Incidence Rate Ratio = 1.10, 95% CI 2-sided [1.02 to 1.18], Standard Deviation 0.05

3. Secondary Outcome: Completion of 9 Month Measles-mumps-rubella Vaccination on Time.
Description: Assess whether patients randomized to the intervention were more likely to have children receiving the measles-mumps-rubella vaccination at 9 months of age after receiving concentrated postpartum counseling compared to women receiving standard of care.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Counseling Existing Providers | Counseling, Retrained Provider
Number analyzed (Participants) | 353 | 344
participants | 211 | 235
Statistical Analysis 1: Comparison: Counseling Existing Providers vs Counseling, Retrained Provider; Test type: Superiority or Other; p = 0.05, Regression, Logistic; The crude analysis result is provided as the odds ratio did not change substantially when adjusted for possible confounders; Odds Ratio (OR) = 1.13, 95% CI 2-sided [1.01 to 1.25], Standard Deviation 0.05

ADVERSE EVENTS:
Arm/Group | Counseling Existing Providers | Counseling, Retrained Provider
Serious Adverse Events (participants affected / at risk) | 0/422 | 0/422
Other Adverse Events (participants affected / at risk) | 0/422 | 0/422

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No